CLINICAL TRIAL: NCT00422201
Title: Prospective, Open-Label, Multicenter, International Study of Mifepristone for Symptomatic Treatment of Cushing's Syndrome Caused by Ectopic Adrenal Corticotrophin Hormone (ACTH) Secretion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070008; 07-CH-0008
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Cushing's Syndrome
Keywords: Cortisol; Cushing's Syndrome; Ectopic ACTH Secretion; Cushing Syndrome
MeSH Terms: conditions — Cushing Syndrome; ACTH Syndrome, Ectopic | interventions — Mifepristone

ARMS (1):
- Prospective, open-label, study of mifepristone (Experimental): Eligible subjects will start study treatment at the dose of 600 mg/day (given as one 200 mg tablet tid, per os). Total duration of treatment will not exceed 12 months. At the end of 12-month treatment, investigators may petition to extend treatment on a case-by-case basis.
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Singe dose

SUMMARY:
This study will evaluate whether the drug mifepristone can improve the symptoms of Cushing's syndrome in people with ectopic adrenal corticotrophin hormone (ACTH) secretion. Cushing's syndrome occurs when the adrenal glands produce too much cortisol, a hormone that helps to regulate the body's use of salt and food. Excessive cortisol is usually the result of too much ACTH, the hormone that causes the adrenal glands to make cortisol. The extra ACTH is made either by a tumor in the pituitary gland (called Cushing's disease) or by a tumor somewhere else (called ectopic ACTH secretion). Mifepristone blocks the action of cortisol in the body. The drug has been used safely to treat a few people with Cushing's syndrome and patients with certain kinds of cancer, gynecological diseases and psychiatric disorders.

People between 18 and 85 years of age with Cushing's syndrome caused by EXCESS ACTH secretion may be eligible for this study. Candidates are admitted to the hospital for evaluation to confirm Cushing's syndrome and to determine its cause. The evaluation includes blood and urine tests, imaging tests, dexamethasone and corticotropin-releasing hormone tests and inferior petrosal sinus sampling. Patients determined to have Cushing's syndrome due to ECTOPIC ACTH secretion undergo imaging studies (CT, MRI and a nuclear medicine scan) and begin mifepristone therapy.

Participants remain in the hospital for the following tests and procedures:

* Physical examination, electrocardiogram (EKG) and blood and urine tests
* Completion of medical questionnaires
* DEXA scan to determine bone mineral density and body composition
* Glucose tolerance test
* Urine pregnancy test and ultrasound to measure uterine lining thickness (for women)

Patients take mifepristone by mouth 3 times a day. The dose is increased every week or so until symptoms improve or the highest dosage allowed is reached. Patients may remain in the hospital for all or part of the dose-finding part of the study. During this period (usually 2 to 4 weeks), blood pressure, glucose tolerance and blood chemistries are measured and EKG and urinalysis done every 5 to 14 days. When the mifepristone dose is stable patients remain on that dose for at least 2 weeks and are then re-evaluated. Patients then return to the hospital for evaluations every 3 months. Those who do well on the drug may continue to take it for up to 12 months.

DETAILED DESCRIPTION:
Between 10% and 20% of patients with hypercortisolism (Cushing's Syndrome) have tumoral ectopic production of adrenocorticotropin hormone (ACTH) that causes cortisol excess. If an ectopic tumor cannot be found or if surgery cannot be done, the treatment options include medicines that reduce cortisol production and bilateral adrenalectomy. The available medications that reduce cortisol production have important adverse effects and are not effective in some patients and adrenalectomy leads to lifelong requirements for medical hormone replacement. Thus, additional treatment options would be welcome. This study evaluates a potential new medication for the treatment of these patients; mifepristone blocks the effects of cortisol rather than decreasing its production. The purpose of this study is to see whether this agent can improve diabetes or other symptoms of Cushing's syndrome in subjects with ectopic ACTH secretion. Another purpose is to evaluate adverse effects with this drug. Patients with presumed ectopic ACTH secretion and diabetes will take mifepristone 600 mg daily by mouth, and the effect on diabetes and other symptoms of Cushing's syndrome will be measured. Subjects will return to the hospital at 2, 3, 6, 9, and 12 months after starting mifepristione for evaluation of diabetes and other symptoms. The agent will be available for up to 12 months for patients in whom it is effective.

Patients take mifepristone by mouth 3 times a day. Each dose will contain 200 mg. Patients may remain in the hospital for all or part of the initial safety studies, every two weeks for eight weeks. During this period blood pressure, glucose tolerance and blood chemistries are measured and EKG and urinalysis done every two weeks. The mifepristone dose can be decreased or stopped if there are adverse effects. When the mifepristone dose is stable for eight weeks, patients will be re-evaluated. Patients then return to the hospital for evaluations one month later and then every 3 months. Those who do well on the drug may continue to take it for up to 12 months.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be included if they have ALL of the three following criteria:

1. Hypercortisolism from Cushing's syndrome caused by ACTH ectopic secretion

   AND
2. Glycemic disorder that is considered to be caused or worsened by the hypercortisolism

   AND
3. At least one symptom attributable to the Cushing's syndrome.

   EXCLUSION CRITERIA:
   * Evidence for Cushing's disease as judged by positive inferior petrosal sinus sampling or a lesion on pituitary MRI with positive CRH test
   * Suspected or known adrenocortical cancer or adenomas, as judged by ACTH values less than 10 pg/ml and adrenal mass
   * Subjects with cyclic Cushing's syndrome defined by any measurement of Urinary Free Cortisol over the previous 2 months less than 2 N
   * Children (age less than 18) and patients over 85 years
   * Pregnant or lactating women. A urinary pregnancy test will be performed in women of childbearing potential unless they have a history of menopause prior to Cushing's syndrome or hysterectomy
   * Life expectancy less than two months
   * Surgery planned within 8 weeks after inclusion, especially bilateral adrenalectomy
   * Uncontrolled diabetes (plasma glucose greater than 15.0 mmol/L (270 mg/L) and/or HbA1c greater than 10%)
   * Uncontrolled hypertension (blood pressure greater than 180/110 mmHg)
   * Recent (less than two weeks prior to inclusion) initiation of corrective treatments for depression
   * Clinically significantly impaired cardiovascular function (e.g. stage IV cardiac failure)
   * Severe liver disease (liver enzymes greater than or equal to 3 x the institutional upper limit of normal range)
   * Severe renal impairment (serum creatinine greater than or equal to 2.2 mg/dl or creatinine clearance less than 30 ml/min)
   * Severe hypokalemia (plasma K below 3.0 mmol/L)
   * Uncontrolled severe active infection
   * In women, known endometrial cancer, history of endometrial hyperplasia or vaginal bleeding of unknown cause
   * Premenopausal women with hemorrhagic disorders or on anticoagulants
   * Recent (less than two weeks prior to inclusion) initiation of or significant change in dose of anti-tumor therapy
   * Previous treatment with approved or experimental steroidogenesis inhibitors, somatostatin analogues within one week of admission (eight weeks for patients on octreotide LAR or on lanreotide autogel)
   * Plasma mitotane concentration greater than 5 microgram/ml
   * Impaired mental capacity or markedly abnormal psychiatric evaluation that precludes informed consent
   * Body weight over 136 kg, which is the limit for the tables used in the scanning areas
   * Inherited porphyria
   * Positive pregnancy test at inclusion
   * Use of antiretroviral agents, midazolam, cabergoline, erythromycin, or grapefruit juice within two weeks of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05-15 (Actual); Primary Completion 2012-04-04 (Actual); Study Completion 2012-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (15):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- France (7):
  - CHU de Bordeaux Hopital Haut Leveque, Bordeaux
  - C.H.U Albert Michallon, Grenoble
  - C.H.U. de Bicetre, Le Kremlin-Bicêtre
  - CHRU de Lille, Lille
  - Hopital de la Timone, Marseille
  - AP-HP, Hopital Cochin Pavillon CORNIL, Paris
  - CHU de Toulouse, Toulouse
- University of Wuerzburg, Wuerzbug, Germany
- Italy (3):
  - Universita Degli Studi, Napoli
  - University of Turin, Orbassano
  - University of Padova, Padua
- Netherlands (3):
  - Internal Medicine Endocrinology, Eindhoven
  - University Hosiptal of Groningen, Groningen
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Background] Bertagna X, Basin C, Picard F, Varet B, Bertagna C, Hucher M, Luton JP. Peripheral antiglucocorticoid action of RU 486 in man. Clin Endocrinol (Oxf). 1988 May;28(5):537-41. doi: 10.1111/j.1365-2265.1988.tb03688.x. PMID 3214945
- [Background] Bertagna X, Escourolle H, Pinquier JL, Coste J, Raux-Demay MC, Perles P, Silvestre L, Luton JP, Strauch G. Administration of RU 486 for 8 days in normal volunteers: antiglucocorticoid effect with no evidence of peripheral cortisol deprivation. J Clin Endocrinol Metab. 1994 Feb;78(2):375-80. doi: 10.1210/jcem.78.2.8106625.
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-CH-0008.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 patients recruited. Recruitment terminated.
Groups:
- Single Arm Mifepristone: Study medication was to be administered at a total daily dose of 600 mg (given as one 200 mg tablet tid, per os) starting on the day of inclusion.
  This dose was to be maintained during the whole study except in case of suspicion of adrenal insufficiency, in which case the dose was temporally stopped for 2 to 3 days and restarted at a lower dose of 400 mg daily until the end of the study.
Period: Overall Study
Arm/Group | Single Arm Mifepristone
Started | 18
Completed | 7
Not Completed | 11

BASELINE CHARACTERISTICS:
Groups:
- Mifepristone: Single arm. Study medication was to be administered at a total daily dose of 600 mg (given as one 200 mg tablet tid, per os) starting on the day of inclusion.
  This dose was to be maintained during the whole study except in case of suspicion of adrenal insufficiency, in which case the dose was temporally stopped for 2 to 3 days and restarted at a lower dose of 400 mg daily until the end of the study.
Arm/Group | Mifepristone
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Region of Enrollment [Number; unit: participants]
  France | 2
  United States | 7
  Netherlands | 6
  Germany | 1
  Italy | 2

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Disorders Improved or Normalized
Description: Criteria for improvement or normalization of glycemic disorders:
  A. For diabetic patients (known or diagnosed at pre-inclusion visit)
  * Decrease in HbA1c > 0.3% B. For patients with IGT
  * Normalization of OGTT (2-hour glucose plasma level after 75 g OGTT < 7.8 mmol/L (140 mg/dL) D. For patients with IFG
  If impaired fasting glucose is also associated with impaired glucose tolerance during OGTT at pre-inclusion:
  - Normalization of OGTT (2-hour glucose plasma level after 75 g OGTT < 7.8 mmol/L (140 mg/dL)
  If impaired fasting glycemia is associated with normal OGTT at pre-inclusion (except at T0):
  - Normalization of fasting plasma glucose (fasting plasma glucose < 5.5 mmol/L (100 mg/dL)
Time Frame: 8 weeks at steady dose
Population: 18 patients were recruited. 7 completed the study but only 3 according to the last protocol version (in which primary efficacy criteria were changed), so only these 3 patients were to be analysed
Measure: Number; unit: participants
Groups:
- Mifepristone: Single arm. Study medication was administered at a total daily dose of 600 mg (given as one 200 mg tablet tid, per os) starting on the day of inclusion.
  This dose was to be maintained during the whole study except in case of suspicion of adrenal insufficiency, in which case the dose was temporally stopped for 2 to 3 days and restarted at a lower dose of 400 mg daily until the end of the study.
Arm/Group | Mifepristone
Number analyzed (Participants) | 3
participants | 2

2. Secondary Outcome: Features of Cushing's Syndrome
Description: Criteria for secondary glycemic disorder improvement of clinical symptoms attributable to the Cushing's syndrome A. For diabetic patients
  * Improvement of the following parameters: glycemic profile, fasting blood glucose, fructosamine, 2-hour OGTT (for diabetics diagnosed at screening)
  * Number of anti-diabetics treatment or dose of anti-diabetics treatment for diabetic patients already on diabetes treatment at inclusion
  * Doses of insulin for insulin-treated patients B. For patients with IGT
  * HbA1c
  * Fructosamine C. For patients with IFG
  * HbA1c
  * Fructosamine D. For all patients
  * Fasting plasma insulin
  * Area Under the Curve of OGTT results when OGTT performed
  * HOMA index
Time Frame: 8 weeks at steady dose
Population: 18 patients were recruited. 7 completed the study but only 3 according to the last protocol version, so only these 3 patients were to be analysed
Measure: Number; unit: participants
Arm/Group | Prospective, Open-label, Study of Mifepristone
Number analyzed (Participants) | 3
participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to the end of the study ie up to 12 months.
Description: Number of patients at risk corresponds to the number of patients who have received study treatment. Among the 18 patients enrolled, 17 received study treament and are considered in the set of population at risk.
Arm/Group | Mifepristone
Serious Adverse Events (participants affected / at risk) | 9/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=17)
Renal acute failure (Renal and urinary disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (2)
Pneumocystis jiroveci (Infections and infestations) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Oedema (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=17)
Nausea (Gastrointestinal disorders) | 7 (30)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (29)
Decreased apetite (Metabolism and nutrition disorders) | 4 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (3)
Dehydratation (Metabolism and nutrition disorders) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 4 (11)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Parotitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sputum purulent (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Adrenal insuffisiency (Endocrine disorders) | 6 (14)
Steroid withdrawal syndrome (Endocrine disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Fatigue (General disorders) | 7 (21)
Pyrexia (General disorders) | 3 (5)
Oedema peripheral (General disorders) | 2 (4)
Oedema (General disorders) | 2 (2)
pain (General disorders) | 1 (1)
C-reactive protein increased (Investigations) | 3 (3)
Blood creatinine increased (Investigations) | 2 (3)
Protein total decrased (Investigations) | 2 (2)
Blood albumin decreased (Investigations) | 1 (2)
Blood corticotrophin increased (Investigations) | 1 (2)
Blood cortisol increased (Investigations) | 1 (2)
Blood urea increased (Investigations) | 1 (2)
High density lipoprotein decreased (Investigations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Cortisol free urine (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1)
Osteocalcin increased (Investigations) | 1 (1)
Proteinuria (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
urine potassium increased (Investigations) | 1 (1)
urine sodium increased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Microalbuminuria (Renal and urinary disorders) | 1 (3)
Nocturia (Renal and urinary disorders) | 1 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Micturition frequency increased (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (25)
Tremor (Nervous system disorders) | 2 (2)
Ageusia (Nervous system disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
As a consequence of the premature study end, analyses performed were primarily descriptive due to the reduced number of enrolled and completed patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less